CLINICAL TRIAL: NCT00801632
Title: Renal Allograft Tolerance Through Mixed Chimerism
Brief Title: Combined Kidney and Bone Marrow Transplantation to Prevent Kidney Transplant Rejection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ITN036ST
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Kidney Transplantation; Kidney Failure, Chronic
Keywords: renal allograft tolerance; mixed chimerism; kidney transplant; bone marrow transplant; antirejection; immunosuppression
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Kidney Transplantation; Bone Marrow Transplantation; siplizumab; Cyclophosphamide; Rituximab; Tacrolimus; Adrenal Cortex Hormones; Methylprednisolone; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Kidney and Marrow Recipients (Experimental): Combined kidney and bone marrow transplant
  Interventions: Procedure: Kidney Transplantation; Procedure: Bone marrow transplantation; Biological: MEDI-507; Drug: cyclophosphamide; Biological: rituximab; Drug: Tacrolimus; Drug: corticosteroids; Radiation: thymic irradiation

INTERVENTIONS:
Procedure: Kidney Transplantation — Surgical transplantation of donor kidney
  Other Names: Renal Transplantation
Procedure: Bone marrow transplantation — During kidney transplant, bone marrow cells donated by the same donor as the kidney are given through a plastic tube placed in a vein in the chest, underneath the collarbone
Biological: MEDI-507 — 0.1 mg/kg on day -2; 0.6 mg/kg on days -1,0,1
  Other Names: siplizumab; anti-CD2 monoclonal antibody
Drug: cyclophosphamide — 60 mg/kg infusion on days -5, -4
  Other Names: Cytoxan
Biological: rituximab — 375 mg/m^2 infusion on days -7, -2, 5, and 12
  Other Names: Rituxan
Drug: Tacrolimus — 0.05 mg/kg intravenously twice daily starting on day -1, adjusted to trough level of 10-15ng/ml, then tapered (if eligible) on days 1, 7, 14, 21, 28, 42, and 56
  Other Names: PROGRAF®
Drug: corticosteroids — 2 mg/kg prednisone on day 4, with an additional 500-mg pulse of methylprednisolone given on days 10, 11, and 12, and then tapered off by day 20
  Other Names: methylprednisolone; prednisone
Radiation: thymic irradiation — 700 cGy of thymic irradiation administered in a single dose on day -1

SUMMARY:
In small initial studies, combined kidney and bone marrow transplants from the same donor have permitted some individuals to stop taking anti-rejection medicines without rejecting their transplant. This clinical trial will study this method in a greater number of people to determine if it is indeed effective and safe.

DETAILED DESCRIPTION:
All patients receiving an organ or tissue transplant must take special medicines known as "immunosuppressive drugs" in order to prevent the immune system from rejecting the transplant. These drugs can be very effective, but they leave the patient at an increased risk of serious infections and certain types of cancer. New methods of preventing transplant rejection are needed.

Researchers have found that transplanting both bone marrow and a kidney from the same donor can create what is called "mixed chimerism." This means that the transplant recipient has a mixture of the donor and recipient's immune systems. It is believed that this mixture of immune cells can prevent rejection of the kidney. In a small prior study, performing a kidney transplant together with a bone marrow transplant from the same donor allowed 4 of 5 patients to stop taking immunosuppressive drugs altogether, without rejecting their transplant. This clinical trial will study more patients to confirm if the technique is safe and effective.

Patients eligible for this study must be candidates for a living kidney transplant, and have an eligible donor identified. The transplant recipient and donor must both consent to participate in this study. Transplant recipients enrolled in the study will receive both kidney and bone marrow transplants from the same living donor. Prior to the transplant procedure, the transplant recipient will undergo a "conditioning regimen" that prepares their immune system for the recipient's immune (bone marrow) cells. This conditioning regimen is a combination of chemotherapy, radiation, immunosuppressive drugs and specialized medications called rituximab and MEDI-507. MEDI-507 is an investigational medication that has not been approved by the FDA. After the transplant procedure, transplant recipients will be prescribed steroids for several weeks and immunosuppressive drugs. After 2 months, the dose of the immunosuppressive drugs will slowly be decreased to zero in patients whose immune system and kidney function meet certain criteria.

Transplant recipients enrolled into the study will be hospitalized for 1 week prior to the transplant procedure. After the transplant, patients will remain in the hospital until the doctor feels they are well enough to go home. Recipients will receive approximately monthly checkups over a period of 2 years after transplant, plus a checkup at 2 ½, 3, 3 ½ , 4, and 5 years after transplant. Checkups will include physical exams, and blood and urine tests to assess immune system and kidney function. At four of these checkups, a kidney biopsy will be requested.

Transplant donors enrolled in the study will attend a screening visit, which will include a physical exam, blood tests and chest x-ray. Eligible donors will be admitted to the hospital for 3-5 days, where bone marrow will be collected prior to removal of the kidney. Transplant donors may be asked at a later date to donate additional blood samples for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Awaiting first or second transplant with a living donor or first transplant with a cadaveric donor
* For living-donor transplants, must have one or more HLA antigen-mismatched donors identified
* Serologic evidence of prior exposure to Epstein-Barr virus (EBV)

Exclusion Criteria:

* ABO blood group-incompatibility for a kidney graft of tissue from a donor
* Decreased circulating white blood cell count
* Positive for HIV-1, hepatitis B and C viruses
* Have had prior radiation therapy that could limit dose
* Lung capacity <50% of predicted normal
* Evidence of insufficient cardiac capacity
* Unwilling to use adequate contraception until 2 years after transplant
* Lactation or pregnancy
* Presence of antibody against the donor

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2008-12; Primary Completion 2014-04 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Sachs, MD, Principal Investigator — Massacusetts General Hospital; Ben Cosimi, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Kawai T, Cosimi AB, Spitzer TR, Tolkoff-Rubin N, Suthanthiran M, Saidman SL, Shaffer J, Preffer FI, Ding R, Sharma V, Fishman JA, Dey B, Ko DS, Hertl M, Goes NB, Wong W, Williams WW Jr, Colvin RB, Sykes M, Sachs DH. HLA-mismatched renal transplantation without maintenance immunosuppression. N Engl J Med. 2008 Jan 24;358(4):353-61. doi: 10.1056/NEJMoa071074. PMID 18216355
- [Result] Kawai T, Sachs DH, Sykes M, Cosimi AB; Immune Tolerance Network. HLA-mismatched renal transplantation without maintenance immunosuppression. N Engl J Med. 2013 May 9;368(19):1850-2. doi: 10.1056/NEJMc1213779. No abstract available. PMID 23656665
- See also: Immune Tolerance Network — http://www.immunetolerance.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with end-stage renal disease and no evidence of prior sensitization were enrolled between December 2008 and September 2009.
Groups:
- MEDI-507: Recipients received a conditioning treatment that started with rituximab (375 mg/m^2 infusion) on days -7, -2, 5 and 12. Cyclophosphamide (60 mg/kg) on days -5 and -4, followed by hemodialysis. MEDI-507, a T-cell-depleting agent, was given at 0.1 mg/kg on day -2 and 0.6 mg/kg on days -1, 0 and 1. Thymic irradiation (700 cGy) was given on day -1. Recipients underwent surgical transplantation of a donor kidney on day 0. During kidney transplant, bone marrow cells donated by the same donor as the kidney were given through a plastic tube placed in a vein in the chest, underneath the collarbone. Prednisone was started at 2 mg/kg/day on day 4 and tapered off by day 20. A steroid pulse (methylprednisolone 500 mg) was given on days 10, 11, and 12. Tacrolimus (0.05 mg/kg twice a day, adjusted to trough level of 10-15 ng/mL) was given starting on day -1. When the subject met weaning criteria, tacrolimus was tapered over a period of no less than 8 weeks beginning 60 days post-transplant.
Period: Overall Study
Arm/Group | MEDI-507
Started | 5
Completed | 4
Not Completed | 1
Not completed — Re-transplant | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat
Arm/Group | MEDI-507
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5
Baseline Creatinine Level [Mean (Standard Deviation); unit: mg/dL] — Baseline creatinine is defined as the lowest serum creatinine collected during the stabilization period or in the 4 weeks following the end of the stabilization period. The stabilization period is defined as 4 consecutive creatinine values close in value (not differing more than 0.3). A normal result is 0.7 to 1.3 mg/dL for men and 0.6 to 1.1 mg/dL for women. Higher results indicate poorer kidney function, as creatinine is removed from the body by the kidneys.
  mg/dL | 1.9 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Successfully Withdrawn Off of Immunosuppressant Medication for 104 Weeks
Description: A participant was considered a success if they were off immunosuppressive therapy for 104 consecutive weeks leading up to study week 208 (48 months post-transplant) or study termination, whichever occurred first.
Time Frame: 48 months post-transplant
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | MEDI-507
Number analyzed (Participants) | 5
participants | 3
Statistical Analysis 1: Comparison: MEDI-507; Test type: Superiority or Other; Percentage of Participants = 60.0, 95% CI 2-sided [14.7 to 94.7] — Clopper-Pearson used to derive confidence interval

2. Secondary Outcome: Percentage of Participants Experiencing Acute Rejection
Description: The percentage of participants who experience an acute rejection. Acute rejection is defined as a biopsy with findings of Banff score of grade IA or higher. The Banff classification is as follows: grade IA is >25% of parenchyma affected and foci of moderate tubulitis; Grade IB is >25% of parenchyma affected and foci of severe tubulitis; Grade IIA is mild to moderate intimal arteritis; Grade IIB is severe intimal arteritis comprising >25% of the luminal area; Grade III is "transmural" arteritis and/or arterial fibrinoid change and necrosis of medial smooth muscle cells with accompanying lymphocytic inflammation.
Time Frame: Transplantation until study completion or participant termination (up to five years)
Population: Intent-to-treat
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MEDI-507
Number analyzed (Participants) | 5
Percentage of Participants | 40 [5.3 to 85.3]

3. Secondary Outcome: Change in Renal Function
Description: Change in renal function as seen in serum creatinine values from baseline until study completion or participant termination. Baseline is defined as the lowest serum creatinine collected during stabilization period or in the four weeks following the end of the stabilization period. The stabilization period is defined as four consecutive creatinine values close in value (not differing more than 0.3 mg/dL). Higher results indicate poorer kidney function, as creatinine is removed from the body by the kidneys.
Time Frame: Transplantation until study completion or participant termination (up to five years)
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MEDI-507
Number analyzed (Participants) | 5
mg/dL
  Baseline Serum Creatinine | 1.9 (1.2)
  Study Termination/Completion | 3.2 (2.7)
  Change from Baseline | 1.2 (1.9)
Statistical Analysis 1: Comparison: MEDI-507; Test type: Superiority or Other; p = 0.215, t-test, 2 sided — P-value based on a paired t-test comparing baseline creatinine level with the level at study completion/participant termination; The test describes whether the average of the difference is different from zero

4. Secondary Outcome: Percentage of Participants With Graft Survival Through 156 Weeks
Description: The percentage of participants with graft survival from transplantation through 156 weeks. Participants who terminated from the study prior to Week 156 without meeting the event were excluded. Graft survival is defined as the time to week 156 or graft loss. Graft loss is defined as the day on which a graft is deemed irreversibly nonfunctional and dialysis is begun, a transplantectomy is performed, or the participant is re-transplanted, whichever comes first. Six consecutive weeks of dialysis are required for the diagnosis of graft loss, though the date of graft loss will be defined as the date of first dialysis.
Time Frame: Transplantation until week 156
Population: Participants who were followed at least three years after transplantation or experienced graft loss prior to week 156
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MEDI-507
Number analyzed (Participants) | 5
Percentage of Participants | 80 [28.4 to 99.5]

5. Secondary Outcome: Percentage of Participants Surviving Through 156 Weeks
Description: The percentage of participants who survived from transplantation through 156 weeks. Participants who terminated from the study prior to Week 156 without meeting the event were excluded.
Time Frame: Transplantation until week 156
Population: Participants who were followed at least three years after transplantation or experienced death prior to week 156
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MEDI-507
Number analyzed (Participants) | 4
Percentage of Participants | 100 [39.8 to 100.0]

6. Secondary Outcome: Time to Neutrophil Recovery Following Transplant
Description: Time (in days) until neutrophil recovery following transplant. Neutrophil recovery is defined as an absolute neutrophil count (ANC) > 500/mm^3 at three consecutive assessments on different days post-transplant. Time to recovery is time from transplantation until the first assessment date used to confirm the recovery.
Time Frame: Transplantation until study completion or participant termination (participants followed up to five years)
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: days
Arm/Group | MEDI-507
Number analyzed (Participants) | 5
days | 14.0 (4.1)

7. Secondary Outcome: Time to Platelet Recovery Following Transplant
Description: Time (in days) until platelet recovery following transplant. Platelet recovery is defined as a platelet count >20,000 /mm^3 and where no transfusion is required. Time to recovery is time from transplantation until platelet value recovers.
Time Frame: Transplantation until study completion or participant termination (participants followed up to five years)
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: days
Arm/Group | MEDI-507
Number analyzed (Participants) | 5
days | 1.0 (0.0)

8. Secondary Outcome: Percentage of Participants Experiencing a Clinically Significant Invasive or Resistant Opportunistic Infection
Description: Clinically significant invasive or resistant opportunistic infections include cytomegalovirus, herpes zoster, and candida.
Time Frame: Transplantation until study completion or participant termination (participants followed up to five years)
Population: Intent-to-treat
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MEDI-507
Number analyzed (Participants) | 5
Percentage of Participants | 0 [0.0 to 52.2]

ADVERSE EVENTS:
Time Frame: Transplantation until study completion or participant termination (up to five years)
Arm/Group | MEDI-507
Serious Adverse Events (participants affected / at risk) | 5/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI-507 (N=5)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Engraftment syndrome (Immune system disorders) | 5 (5)
Transplant rejection (Immune system disorders) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI-507 (N=5)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Catheter related complication (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (4)
Drug toxicity (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Weight increased (Investigations) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 4 (4)
Renal failure acute (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No